CLINICAL TRIAL: NCT03017248
Title: Benefit of the Association of Low Doses of Ketamine With Intravenous Morphine in the Treatment of Acute Severe Pain in Emergency Department
Brief Title: Low-dose Ketamine for Acute Pain in the Emergency Department
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, HAJER KRAIEM, M.D, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMSousse
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Pain
Keywords: pain; ketamine; morphine; analgesia; emergency
MeSH Terms: conditions — Pain; Agnosia; Emergencies | interventions — Ketamine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Morphine and Placebo (Active Comparator): Morphine IV, Dose: 0.1 mg/Kg followed 10 minutes later by an injection of Placebos (0.9% normal saline 0.05ml/kg)
  Interventions: Drug: Placebos; Drug: Morphine
- Morphine and Ketamine 0.15 (Experimental): Morphine IV, Dose: 0.1 mg/Kg followed 10 minutes later by an IV bolus of Ketamine at the dose of 0.15mg/kg
  Interventions: Drug: Ketamine; Drug: Morphine
- Morphine and Ketamine 0.3 (Experimental): Morphine IV, Dose: 0.1 mg/Kg followed 10 minutes later by an IV bolus of Ketamine at the dose of 0.3mg/kg
  Interventions: Drug: Ketamine; Drug: Morphine

INTERVENTIONS:
Drug: Ketamine — ketamine
  Other Names: Ketalar, 50 Mg/mL Injectable Solution
  Arms: Morphine and Ketamine 0.15; Morphine and Ketamine 0.3
Drug: Placebos — 0.9% normal saline
  Other Names: Normal Saline Flush, 0.9% Injectable Solution
  Arms: Morphine and Placebo
Drug: Morphine — Morphine
  Other Names: Morphine Sulfate

SUMMARY:
This study aims to determine the efficacy and safety of low dose ketamine in association with IV morphine in the management of acute moderate to severe pain in emergency department.

The investigators hypothesize that low dose ketamine will result in more effective pain control than morphine alone and will not be associated with an increase in adverse events.

DETAILED DESCRIPTION:
Management of pain in the Emergency Department is challenging. Treatment of pain is most often accomplished by parenteral opioids analgesics. However, the use of opioids alone for pain control is often associated with inadequate analgesia and increased adverse events.

Low-dose ketamine has been shown to improve pain perception and produce an opioid-sparing effect when given perioperatively.

Its use in the ED may probably play a role in maximizing analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give informed consent
* Comfortable with the experimental protocol as outlined to them by the research team
* Severe pain, pain score of at least 50/100 on Visual Analogue Scale (VAS) or 5/10 numerical ratings score
* Acute pain, pain duration < 7days
* Deemed by treating ED attending physician to require IV opioid analgesia

Exclusion Criteria:

* Neurologic, respiratory, or hemodynamic compromise
* Pregnancy or breastfeeding
* Known or suspected allergy to ketamine or morphine
* Known Renal (Cr>2.0) or Liver Failure
* Unstable psychiatric disease (as per treating physician)
* History of stroke
* History of cardiac disease or coronary artery disease
* History of chronic respiratory disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of analgesia: To assess the primary outcome of pain relief, we used patient-reported pain scores. We consider the pain decreasing of at least 50% of pain score and the summed pain-intensity difference (SPID) over 2 hours | Two hours after starting protocol
  At baseline, to assess our primary aim, efficacy of pain control, we will use patient reported pain scores and amount of rescue analgesia (parenteral morphine) received. Trained residents will ask participants to report their pains scores using a numerical pain rating scale (NPRS). The NPRS used will be a 0 to 10 rating scale. Baseline NPRS will be measured after randomization, but just before administration of morphine. Change in reported pain score during the protocol will be analysed.
  The SPID was calculated using the pain-intensity difference (PID) at each of these study time points. The PID for a given time point is equal to the baseline NPRS minus the subsequent NPRS at each study time point. SPID is the summation of the PID at each of the study time points, weighted using the amount of time since the prior assessment

SECONDARY OUTCOMES:
Total patient-perceived pain relief | Two hours after starting protocol
  The total patient-perceived pain relief will be calculated using weighted sum of the pain relief scale performed at each study time point. This pain relief scale is a five-point scale that asks participants to rate pain relief as complete = 4, a lot = 3, some = 2, a little = 1, and none = 0
Amount of rescue analgesia received | Two hours after starting protocol
  The amount of rescue analgesia received (in milligrams of morphine equivalents) will be recorded.
Time to rescue analgesia | Two hours after starting protocol
  Time to rescue analgesia will be calculated as the time from administration of the last study medication (placebo or ketamine) to administration of an opioid analgesic.
The occurrence of adverse events | Two hours after starting protocol
  We will record participant-reported dizziness, nausea, vomiting, confusion, dysphoria, visual disturbances, or other complaints at baseline and each study time point. All patients will be monitored for the duration of the study period and vital signs will be recorded at each time point.
  The presence of tachycardia (heart rate > 100 beats/min.), hypotension (systolic blood pressure [sBP] < 100 mm Hg), hypertension (sBP > 180 mm Hg or diastolic blood pressure [dBP] > 100 mm Hg), and respiratory depression (respiratory rate < 12 breaths/min, oxygen saturation < 92%, or need for supplemental oxygen) will be noted.
The total dose of morphine administered | Two hours after starting protocol
  The amount of rescue analgesia will be recorded at each time point and the total dose calculated

CONTACTS AND LOCATIONS:
Overall Officials: Hajer KRAIEM, MD, Principal Investigator — Faculty of medicine of Sousse
Locations (1):
- Faculty of medicine of Sousse, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided